CLINICAL TRIAL: NCT01979055
Title: Use of a Self-regulation Intervention to Improve Control and Outcomes in Older Adults With Asthma
Brief Title: Achieving Better Control for Older Adults With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Alan Baptist, MD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00076471
Record Dates: First submitted 2013-10-28; First posted 2013-11-08 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Asthma; Elderly
Keywords: asthma; older adults; elderly; behavior
MeSH Terms: conditions — Asthma; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-regulation intervention (Experimental): 6 session educational intervention (3 telephone, 3 In-person), led by a health educator
  Interventions: Behavioral: Self-regulation intervention
- Control group (Placebo Comparator): 3 telephone calls to assess any additional questions regarding asthma
  Interventions: Behavioral: Telephone follow-up

INTERVENTIONS:
Behavioral: Self-regulation intervention — 6 session educational intervention (3 telephone, 3 In-person), led by a health educator
  Arms: Self-regulation intervention
Behavioral: Telephone follow-up — Usual care group, will also receive 3 telephone calls to assess any questions they may have about asthma
  Arms: Control group

SUMMARY:
Asthma in older adults has been overlooked, understudied, and inadequately treated. While asthma programs targeting the unique needs of children, teenagers, women, minorities, and other populations have been successfully developed, there are currently none for older adults. This is particularly distressing as the asthma hospitalization rates, mortality rates, quality of life, and control are significantly worse in the elderly as compared to other age groups. It is clear that novel approaches are needed to improve the care in this population.

The investigators group has been active in the research of asthma in the elderly. The investigators have analyzed national asthma data sets to look for disparities in older adults, have conducted qualitative research to determine factors associated with poor control in the elderly, and have performed a pilot study of a self-regulation intervention which was able to improve outcomes. The investigators also have over 20 years of experience in asthma self-regulation interventions and physician communication enhancement for multiple populations of asthma patients. The investigators will combine these strengths into their current protocol.

The intervention program will be based on the self-regulation theory of behavior, which will enhance the participants' ability to self-manage this chronic condition, actively involve the participant in their own health care management, and produce sustained results. In this proposal, the investigators will evaluate a self-regulation asthma intervention in a diverse population of older adults. The intervention will be personalized to the challenges and goals each individual faces, which will enhance its applicability in different populations. This intervention will incorporate standard asthma education, complementary techniques for which older adults have expressed a strong interest, and enhanced communication with each participant's physician. Asthma specific outcomes will be assessed at 1, 6, and 12 months. The primary goal of this intervention is to decrease health care utilization (emergency department, urgent care, hospital, and unscheduled visits) for older adults with asthma. The investigators will also assess the ability to improve quality of life, asthma symptoms, asthma control, lung function parameters, self-efficacy, and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 55
* persistent asthma,
* have a primary care physician (PCP) who is willing to receive email communication during the study.

Exclusion Criteria:

* any other significant cardiopulmonary disease (including chronic obstructive pulmonary disease)
* a greater than 20 pack-year smoking history
* lack of telephone access
* decreased cognitive capacity such that participation in the program would not be possible

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2013-11; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Health care utilization | 12 months
  Health care utilization (ED visits, hospitalizations, and unscheduled urgent care visits)

SECONDARY OUTCOMES:
Asthma Quality of Life | 12 months
  Asthma Quality of Life Questionnaire (AQLQ)
Asthma control | 12 months
  Asthma Control test (ACT)
Asthma costs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan Baptist, MD, MPH, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan

REFERENCES:
- [Derived] Bennett GH, Carpenter L, Hao W, Song P, Steinberg J, Baptist AP. Risk factors and clinical outcomes associated with fixed airflow obstruction in older adults with asthma. Ann Allergy Asthma Immunol. 2018 Feb;120(2):164-168.e1. doi: 10.1016/j.anai.2017.10.004. Epub 2017 Dec 28. PMID 29290515